CLINICAL TRIAL: NCT03285893
Title: Quantitation of Oral Cell DNA Adducts in Smokers
Brief Title: Oral Cell DNA Adducts in Smokers
Acronym: OCDNA
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: University of Hawaii (Other)
Responsible Party: Sponsor
Other Study IDs: 2017NTLS019
Record Dates: First submitted 2017-09-01; First posted 2017-09-18 (Actual); Results first posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-09

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — oral cell DNA and urine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Native Hawaiian cigarette smokers: oral cell DNA adducts
  Interventions: Other: oral cell DNA adducts
- White (European Americans) cigarette smokers: oral cell DNA adducts
  Interventions: Other: oral cell DNA adducts
- Japanese American cigarette smokers: oral cell DNA adducts
  Interventions: Other: oral cell DNA adducts

INTERVENTIONS:
Other: oral cell DNA adducts — oral cells will be collected, DNA isolated, and analyzed for adducts

SUMMARY:
DNA adducts in the oral mucosa cells of 100 smokers from 3 ethnic groups - Native Hawaiians, Whites, and Japanese Americans with differing risks for lung cancer upon cigarette smoking will be quantified. DNA adducts of tobacco smoke carcinogens will be quantified using both targeted and untargeted approaches.

DETAILED DESCRIPTION:
Using high resolution mass spectrometry, quantify known DNA adducts in oral mucosa cells of 100 smokers from each ethnic group - Native Hawaiians, Whites, and Japanese Americans. DNA adducts of tobacco-specific compounds, formaldehyde, and acrolein will be quantified.

2. Analyze the urine of 100 smokers and 100 non-smokers from each of these groups for mercapturic acids of acrolein and crotonaldehyde, as well as total nicotine equivalents and total NNAL (smokers only). These data will provide critical information relevant to the high risk of Native Hawaiians for lung cancer, and in relationship to the DNA adduct measurements of Specific Aim 1.

ELIGIBILITY:
Inclusion Criteria:

* currently smoke at least 5 cigarettes per day, self-identified Japanese Americans, European Americans, or Native Hawaiians.

Exclusion Criteria:

* no current use of other nicotine containing products, no acute or uncontrolled medical or psychiatric conditions, no greater than 14 alcoholic drinks per week, not pregnant, not breastfeeding, not currently taking any medications that affect relevant metabolic enzymes, no active infection.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 100 each of three ethnic groups: Native Hawaiians, Japanese Americans, whites
Sampling Method: Probability Sample
Enrollment: 281 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stepehn Hecht, PhD, Principal Investigator — University of Minnesota
Locations (1):
- Tobacco Use Research Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided
Only unidentified data will be shared.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Native Hawaiian Cigarette Smokers | White (European Americans) Cigarette Smokers | Japanese American Cigarette Smokers
Started | 101 | 101 | 79
Completed | 101 | 101 | 79
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Native Hawaiian Cigarette Smokers | White (European Americans) Cigarette Smokers | Japanese American Cigarette Smokers | Total
Number analyzed (Participants) | 101 | 101 | 79 | 281
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (17.7) | 47.5 (15.7) | 59.2 (14.6) | 50.1 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 49 | 26 | 128
  Male | 48 | 52 | 53 | 153
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 79 | 79
  Native Hawaiian or Other Pacific Islander | 101 | 0 | 0 | 101
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 101 | 0 | 101
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Concentration of γ-OH-Acr-dGuo, a Major Acrolein-DNA Adduct
Description: Acrolein-DNA adduct (8R/S)-3-(2'-deoxyribos-1'-yl)-5,6,7,8-tetrahy- dro-8-hydroxypyrimido[1,2-a]purine-10(3H)-one. Model adjusted for age, sex and race/ethnicity
Time Frame: Baseline
Measure: Mean (Inter-Quartile Range); unit: 10^9 nucleotides/mL
Arm/Group | Native Hawaiian Cigarette Smokers | White (European Americans) Cigarette Smokers | Japanese American Cigarette Smokers
Number analyzed (Participants) | 101 | 101 | 79
10^9 nucleotides/mL | 49.7 [41.2 to 59.9] | 67.1 [55.7 to 80.7] | 46.5 [37.2 to 58.0]

2. Secondary Outcome: εdAdo, Per 10^9 Nucleotides
Description: Lipid peroxidation-related adduct 1,N6-etheno-dAdo etheno-DNA adducts from peroxidation of lipids. Model adjusted for age, sex and race/ethnicity
Time Frame: Baseline
Measure: Mean (Inter-Quartile Range); unit: 10^9 nucleotides/mL
Arm/Group | Native Hawaiian Cigarette Smokers | White (European Americans) Cigarette Smokers | Japanese American Cigarette Smokers
Number analyzed (Participants) | 101 | 101 | 79
10^9 nucleotides/mL | 11.3 [9.9 to 12.9] | 11.3 [9.94 to 12.9] | 9.16 [7.83 to 10.7]

ADVERSE EVENTS:
Description: No adverse events collected, single visit observational study
Arm/Group | Native Hawaiian Cigarette Smokers | White (European Americans) Cigarette Smokers | Japanese American Cigarette Smokers
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-02): https://cdn.clinicaltrials.gov/large-docs/93/NCT03285893/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-05): https://cdn.clinicaltrials.gov/large-docs/93/NCT03285893/ICF_001.pdf